CLINICAL TRIAL: NCT02113488
Title: Case-control Study: Causes of Nonattendance at Clinical Medicine Scheduled Outpatient Appointments in a University General Hospital
Brief Title: Causes of Nonattendance at Scheduled Outpatient Appointments
Acronym: AU2
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1978
Record Dates: First submitted 2014-04-01; First posted 2014-04-14 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Appointments and Schedules; Outpatient Clinics, Hospital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: P: Patients who did attend a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)
- Case: A: Patients who did not attend (A) a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)
- Control: C: Patients who cancelled (C) a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

SUMMARY:
Our aim was to identify the causes non-attendance at scheduled appointments at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA).

DETAILED DESCRIPTION:
Nonattendance at scheduled appointments at outpatient clinics is a common problem in general medical practice, representing a significant cost to the health care system, and resulting in disruption of daily work planning.Nonattendance at medical appointments has consequences not only for doctors (as it requires a greater use of resources and time), but also for patients, because there may be deterioration in the quality of care, and dissatisfaction associated with delays in obtaining a new appointment.

ELIGIBILITY:
Inclusion Criteria:

* Over 17 years
* Adults who attended, did not attend and cancelled a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

Exclusion Criteria:

* Refusal to register or to the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a scheduled appoitment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Causes of nonattendance | Between the scheduled appointment and 48 hours after
  Patients who did not attend a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

SECONDARY OUTCOMES:
Causes of cancelation | Between the scheduled appointment and 48 hours after
  Patients who cancelled a scheduled appointment at the Clinical Medicine Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires (HIBA)
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Argentina